CLINICAL TRIAL: NCT07061236
Title: The Effect of Education on Comfort and Anxiety Levels in Patients Receiving 5-FU Treatment Administered With an Elastomeric Pump: A Randomized Controlled Trial
Brief Title: Education Effect on Comfort and Anxiety in 5-FU Elastomeric Pump Therapy
Acronym: EDUCAP-5FU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Anita Karaca, Assist. Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AKaraca; AKaraca (Other: BiruniU)
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Comfort; Chemotherapy; Education
Keywords: Anxiety, Cancer, Chemotherapy, Nurses, Port Catheters
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to intervention or control group
Masking Description: No masking was performed due to the nature of the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Patients will receive face-to-face training on the use of the elastomeric pump with 5-FU, supported by an educational booklet.
  Interventions: Other: Elastomeric Pump Education
- Control group (No Intervention): Patients will receive standard institutional care without any additional education or training.

INTERVENTIONS:
Other: Elastomeric Pump Education — This intervention involves a 15-20 minute face-to-face training session about the use of the elastomeric pump with 5-FU, supported by visual materials and an educational booklet developed by the researchers based on current literature and expert opinion
  Arms: Intervention Group

SUMMARY:
Cancer is a chronic disease with an increasing global prevalence and high mortality rates. Surgical interventions, radiotherapy, and especially chemotherapy are among the main treatment modalities. Although chemotherapy prolongs survival, it also causes serious physical and psychological side effects. The prolonged and repetitive nature of chemotherapy necessitates safe vascular access, for which port catheters are frequently preferred. These subcutaneously implanted devices reduce the risk of complications and offer significant advantages in outpatient treatment settings.

5-Fluorouracil (5-FU), commonly used in the treatment of metastatic colorectal cancer, requires prolonged intravenous infusion to be effective. In this context, elastomeric pumps (EPs) are portable, user-friendly, non-electronic medical devices that allow for the continuous and controlled administration of 5-FU. EPs enable patients to continue chemotherapy at home, reducing hospital stays and enhancing both patient satisfaction and quality of life. However, environmental factors such as temperature, viscosity, and gravity may cause variations in flow rate, posing potential safety risks. Therefore, nurses must be competent in the use of EPs, patient education, and management of possible complications.

The use of EPs not only affects treatment efficacy but also has a significant impact on the comfort levels and anxiety of cancer patients. Home-based chemotherapy with EPs helps patients cope with uncertainty, fear, and stress associated with the diagnosis and treatment process. Delivering care outside the hospital environment reduces psychological burden and supports the individual's autonomy and social life. Thus, the wider implementation of EPs in 5-FU treatment and the active involvement of nurses in this process contribute substantially to both treatment outcomes and the overall patient experience. This study was designed to evaluate the impact of education provided to chemotherapy patients receiving 5-FU treatment via elastomeric pumps on their comfort and anxiety levels.

Hypotheses:

H1: There is a significant difference in comfort levels between patients educated about 5-FU treatment administered via elastomeric pumps and those receiving standard education.

H2: There is a significant difference in anxiety levels between patients educated about 5-FU treatment administered via elastomeric pumps and those receiving standard education.

H3: Certain variables have a significant effect on the comfort levels of chemotherapy patients receiving 5-FU treatment via elastomeric pumps.

H4: Certain variables have a significant effect on the anxiety levels of chemotherapy patients receiving 5-FU treatment via elastomeric pumps.

The study will be conducted as a randomized controlled trial. At study initiation, participants in both the intervention and control groups will complete the Patient Information Form, General Comfort Questionnaire-Short Form, Beck Anxiety Inventory, and Informed Consent Form during a face-to-face interview. Participants in the intervention group will additionally receive a 15-20 minute training session on the use of the elastomeric pump with 5-FU, based on a patient education booklet developed from current literature, delivered through verbal explanations and visual materials. The control group will follow standard institutional procedures without supplementary training. Follow-up assessments, including the General Comfort Questionnaire-Short Form and Beck Anxiety Inventory, will be re-administered to all participants during face-to-face interviews one month after baseline.

DETAILED DESCRIPTION:
Cancer is a chronic and fatal disease with an increasing global incidence. According to the 2022 Global Cancer Report prepared by the International Agency for Research on Cancer (IARC), a specialized agency of the World Health Organization, there were approximately 20 million new cancer cases and 10 million cancer-related deaths worldwide. Demographic projections estimate that the number of new cancer cases per year will rise to 35 million by 2050, representing a 77% increase compared to 2022 (International Agency for Research on Cancer [IARC]). Cancer is a progressive disease, and as it advances, patients may experience various physical and psychological symptoms. Many of these symptoms arise not from the disease itself but as side effects of chemotherapy (Temiz and Durna, 2020). Surgical interventions, radiotherapy, and chemotherapy are among the primary treatment methods for cancer. Although chemotherapy positively affects survival, it is also associated with severe physical and psychological side effects. Due to the long-term and repetitive nature of chemotherapy, ensuring safe intravenous administration of chemotherapeutic agents is crucial (Chefchaouni et al., 2023; Burucu and Polat, 2024).

A port catheter is a closed system consisting of a catheter that extends into the central vein, a subdermal reservoir connected to the catheter, and a specialized needle inserted from the dermis into the reservoir (Özden et al., 2012; Paleczny et al., 2013). Typically implanted over the upper pectoral muscle in the upper thoracic region (chest port), port catheters can also be placed in the upper arm or femoral (inguinal) region as alternatives (Paleczny et al., 2013; Pinelli et al., 2018). These subcutaneously implanted vascular access devices facilitate the infusion of chemotherapeutic agents, provide fluid support, and ensure long-term supportive care when needed. They allow for outpatient chemotherapy administration, enabling patients to return home on the same day, thereby increasing patient satisfaction (Burucu and Polat, 2024).

Given the extended duration of cancer treatment, port catheters are preferred over other central venous catheters. Their subcutaneous placement reduces the risk of complications such as occlusion, infection, dislocation, thrombosis, extravasation, phlebitis, and bleeding, and eliminates the need for dressing after wound healing (Odabas et al., 2014; Kesici et al., 2017; Pu Y-L et al., 2020). With specialized knowledge, attention, and experience, port catheters can be used safely for many years (Esfahani et al., 2015; Önder et al., 2014). While implantation is the responsibility of the clinician, needle insertion, catheter care, and initiating appropriate interventions in case of complications require a team effort in which nurses play a central role (Yeşil et al., 2014). Before port needle insertion, nurses inform patients and their families about the rationale for catheter insertion, the procedure, necessary precautions, possible complications, and symptoms. Patients sign an informed consent form. A detailed medical history is obtained, allergies are queried, and premedication is administered if necessary (Oran, 2009; Turan and Cantürk, 2013; Yeşilbalkan, 2005).

Needle access to the port may cause procedural pain and anxiety, reducing patient comfort. Healthcare professionals bear significant responsibility in minimizing these effects (Kutlu, 2015). Physicians and nurses must provide continuous education to patients and families to ensure optimal care (Yeşilbalkan, 2005). Accordingly, nurses' knowledge and experience regarding port catheter care are crucial. Nurses, as vital providers of healthcare, have critical responsibilities in safely performing interventions, preventing and detecting complications early, and educating patients and their families about catheter care (Öztaş et al., 2022). Studies show that informed patients experience less anxiety and fear, whereas uninformed patients are more affected by early-stage complications (Uslu et al., 2019).

5-Fluorouracil (5-FU) remains one of the most commonly used antineoplastic agents for advanced colorectal cancer. To exert its effect, 5-FU must be converted into a nucleotide. As an antimetabolite chemotherapy drug, 5-FU can be administered via intravenous infusion over 5-10 minutes, 20-60 minutes, or as continuous infusions over 22-24 hours for one to four days. Common side effects include bone marrow suppression, nausea, vomiting, anorexia, sore throat, hair loss, and diarrhea. Rare side effects include gait disturbances, eye irritation, confusion, severe allergic reactions, and cardiac complications such as acute coronary syndrome, cardiomyopathy, vasospastic angina, heart failure, arrhythmias, and sudden cardiac death. Cardiac effects usually subside after discontinuation of the infusion (Stewart et al., 2012; Shoemaker et al., 2004).

Elastomeric pumps (EPs) are devices that allow for quantitative and continuous drug delivery without electronic control. They are used to administer antibiotics, analgesics, and antineoplastic agents (Abe et al., 2021). An important advancement in oncology practice has been the gradual shift of chemotherapy to outpatient and home-based settings, optimizing hospital capacity and improving patient satisfaction (Chefchaouni et al., 2023). Regimens such as FOLFOX and FOLFIRI for colorectal cancer and FOLFIRINOX for pancreatic cancer require 46-hour continuous infusions of 5-FU, often delivered via EPs. These devices operate at a fixed flow rate and do not require speed adjustment, making them reliable and safe. The transition from inpatient to outpatient treatment has reduced the burden on patients and increased satisfaction. Even in home care, EPs facilitate continuous drug delivery and are thus widely used (Abe et al., 2021).

EPs have become a preferred treatment method in many chemotherapy regimens due to their cost-effectiveness and reduction in hospital stays, personnel demands, and supply use. However, their safe and effective use depends on offering outpatient chemotherapy to suitable patients. Despite their ease of use, EPs are not risk-free. The cytotoxic nature of the infused drugs means that pump malfunctions may pose significant safety risks. Environmental factors such as temperature, viscosity of the chemotherapy solution, and the height of the EP relative to the catheter can affect flow rate and cause inconsistencies. Thus, the pump accompanying the patient home must be reliable and accurate to ensure comfort and safety. An ideal pump should maintain both high consistency and accuracy in its flow profile (Chefchaouni et al., 2023). Studies on technical failures of EPs are limited, especially regarding outpatient use. For example, Kia et al. (2023) surveyed chemotherapy-related incidents involving EPs, reporting 46 EP-related issues out of 213 events, including pump malfunction and incorrect flow rate (Chefchaouni et al., 2023).

The side effects of cancer treatment negatively affect both patients and their families emotionally, physically, and socioeconomically, lowering their quality of life. Anxiety in response to cancer treatment often goes unrecognized and untreated. Events that may provoke anxiety include hearing the diagnosis, receiving chemotherapy, and discussing family-related issues. Anxiety symptoms are reported in 20-60% of cancer patients. Oncologists often prioritize the treatment of cancer over psychiatric conditions, which may lead to the underdiagnosis of anxiety (Kaykunoğlu and Tambağ, 2022).

A cancer diagnosis, disease symptoms, lack of information, perceived loss of control, uncertainty about treatment efficacy, and prognosis can create psychological distress. Patients may experience anxiety, anger, guilt, hopelessness, helplessness, isolation, fear, and resistance to the illness. Chemotherapy may lead to physical symptoms such as alopecia, nausea, vomiting, and diarrhea, as well as psychological symptoms like anxiety, depression, and anger. These effects may disrupt treatment adherence, compromise coping mechanisms, and impair future expectations. The psychological side effects of chemotherapy, such as fear, depression, and anxiety, adversely impact daily functioning (Hindistan et al., 2015).

In chemotherapy practice, nurses have key responsibilities including educating patients and families, recognizing side effects and toxicities, and ensuring patient engagement. Effective nursing care helps patients cope with the major stressors associated with cancer. Supporting patients in expressing emotions and managing the physical and psychological stress of cancer is vital. Identifying psychological symptoms in chemotherapy patients is essential to support well-being, prevent health issues, enhance self-care, promote positive health behaviors, and provide systematic nursing interventions (Hindistan et al., 2015).

A cancer diagnosis may trigger emotional, psychological, and behavioral responses such as guilt, abandonment, anxiety, pain, grief, and fear of death, all of which can diminish patient comfort and well-being. Common social challenges include isolation, role changes, job loss, interpersonal conflicts, and social withdrawal. Comfort has been defined as the absence of pain, distress, anxiety, and discomfort, and analyzed by Katharina Kolcaba, who described it as the momentary experience of relief, ease, or transcendence in the physical, psychospiritual, environmental, and sociocultural contexts. Patient and family education aims to enhance comfort during disease management. One study found that comfort increased as patients managed chemotherapy symptoms (Can and Hindistan, 2021).

Unmet comfort needs may lead to feelings of threat, loss, uncertainty, limitation, deprivation, and anxiety in cancer patients. Such unmet needs can foster negative expectations for future interventions, reduce self-confidence, and increase anxiety levels (McCarthy et al., 2013). Higher anxiety levels are associated with reduced psychospiritual comfort. Therefore, patients may experience both greater anxiety and lower comfort levels (Yilmaz and Arslan, 2015). Physical, psychospiritual, sociocultural, and environmental comfort levels are closely linked to quality of life. Nursing interventions aimed at increasing comfort in oncology patients can directly influence their quality of life (Kim and Kwon, 2007; Hou et al., 2007). Literature indicates that patient education reduces anxiety, improves coping, and plays a significant role in patient satisfaction (Gürlek and Yavuz, 2013; Sayin and Aksoy, 2012).

Education of patients receiving outpatient 5-FU treatment is essential. EPs have revolutionized home-based chemotherapy, being widely accepted for their reliability, consistency, ease of use, and management. When used as recommended and environmental factors are controlled, they are well-received by the public. Continuous training of healthcare providers and patients helps prevent malfunctions and ensures safe and effective use of EPs (Chefchaouni et al., 2023). For nurses to effectively participate in patient education, they must possess adequate knowledge. Providing comprehensive education before discharge may enhance patient compliance and comfort and reduce anxiety during 5-FU chemotherapy.

Objective: This study was designed to evaluate the impact of education provided to chemotherapy patients receiving 5-FU treatment via elastomeric pumps on their comfort and anxiety levels.

Study Design, Setting, and Sample: This research was planned as a randomized controlled trial. The study is scheduled to be conducted at the Medical Oncology Outpatient Clinic of Koç University Hospital between February and July 2025, following ethical approval from the Koç University Ethics Committee and institutional permission from the relevant hospital.

The study population will consist of chemotherapy patients receiving 5-FU treatment via an elastomeric pump at a foundation university hospital located on the European side of Istanbul, which serves as a tertiary care center. The study will be conducted as a randomized controlled trial.

To determine the required sample size, a power analysis was performed using the G*Power 3.1 software. In a similar study conducted by Silgan (2024), the effect size related to anxiety difference was calculated as 0.740. To achieve a power of at least 95% with a significance level of 5% and an effect size of 0.740, it was determined that 31 patients per group (62 total) are necessary (df=30; t=1.697). Considering the need for high statistical power and potential dropouts, the target sample size was set at 37 patients per group, totaling 74 participants.

In order to avoid bias in the selection of participants for the study, randomization will be applied. The randomization table was created using the website "https://www.calculatorsoup.com".

Inclusion Criteria:

* Diagnosed with cancer,
* Able to understand Turkish and literate,
* Medically fit to participate in the study,
* Willing to participate in the study,
* Aged 18 years or older.

Exclusion Criteria:

* Diagnosed with a psychiatric disorder,
* Unable to communicate effectively,
* Refusing to participate in the study.

Data Collection Instruments:

Data for the study will be collected using the "Patient Information Form," the "General Comfort Questionnaire - Short Form," and the "Beck Anxiety Inventory."

Patient Information Form: This form, prepared by the researcher based on a literature review, consists of two sections: Socio-Demographic Characteristics and Features Related to 5-FU Treatment, comprising a total of 15 questions.

General Comfort Questionnaire - Short Form (GCQ-SF): The GCQ-SF was developed by Kolcaba in 2006. Its Turkish validity and reliability study was conducted by Çıtlık et al. (2018). The GCQ-SF comprises three subdimensions: ease, relaxation, and transcendence. Specifically, the subdimensions include ease (9 items), relaxation (9 items), and overcoming problems (10 items). The scale consists of both positively and negatively worded items; during scoring, negatively worded items are reverse-coded before summation. The total score is then divided by the number of items to obtain a mean score. The lowest possible score of 1 indicates low comfort, whereas the highest score of 6 indicates high comfort. The negatively worded items include items 2, 3, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 21, 23, 24, 25, and 27. The Cronbach's alpha reliability coefficient of the Turkish version of the GCQ-SF was found to be 0.82. The Cronbach's alpha values for the subdimensions ease, relaxation, and transcendence were 0.81, 0.81, and 0.76, respectively (Çıtlık et al., 2018).

Beck Anxiety Inventory (BAI): Developed by Beck et al. (1988), the BAI measures the prevalence of anxiety symptoms experienced by individuals. Its Turkish adaptation was performed by Ulusoy et al. (1998). The self-report scale consists of 21 items, each scored between 0 and 3, with total scores ranging from 0 to 63. Scoring interpretation is as follows: 0 represents no anxiety, 1 mild, 2 moderate, and 3 severe anxiety. Higher total scores indicate greater severity of anxiety symptoms. The scale includes items assessing anxious temperament, autonomic hyperactivity, motor tension, and certain cognitions. Participants are asked to evaluate symptoms experienced "during the past week, including today." Scores between 0-7 indicate minimal or no anxiety, 8-15 mild anxiety, 16-25 moderate anxiety, and 26-63 severe anxiety. Although not definitive, medical treatment is generally recommended for individuals scoring above 16. Treatment decisions should consider both scale scores and clinical evaluation. Ulusoy et al. (1998) reported a Cronbach's alpha of 0.93 for the scale's internal consistency (Ulusoy et al., 1998).

Data Collection Method: The research data will be collected through face-to-face interviews conducted with volunteers participating in the study, using the designated data collection instruments.

Procedures for the Intervention Group: Similarly, patients meeting the inclusion criteria and consenting to participate will sign the Informed Consent Form and complete the Patient Information Form, the Short Form of the General Comfort Questionnaire, and the Beck Anxiety Inventory within approximately 15-20 minutes. Education will then be provided by the researcher based on current literature and the educational materials prepared by the B-Braun brand for the elastomeric pump, supplemented by a specifically prepared training booklet. Patients will be advised to contact the relevant researcher if any issues arise. The education session is expected to last approximately 15 minutes. The effectiveness of the education will be re-evaluated at the end of the first month of the study using the Short Form of the General Comfort Questionnaire and the Beck Anxiety Inventory.

Procedures for the Control Group: Patients who apply to the medical oncology outpatient clinic for 5-FU treatment via elastomeric pump, meet the inclusion criteria, and consent to participate in the study will be asked to sign an Informed Consent Form. Subsequently, they will complete the Patient Information Form, the Short Form of the General Comfort Questionnaire, and the Beck Anxiety Inventory, which will take approximately 15-20 minutes. During the study period, patients will continue to receive routine education, follow-up, and treatment. At the end of the first month of the study, the Short Form of the General Comfort Questionnaire and the Beck Anxiety Inventory will be reassessed.

Data Analysis The data obtained in the study will be analyzed using SPSS for Windows version 22.0. The Kolmogorov-Smirnov test will be used to determine whether the data follow a normal distribution. If the Kolmogorov-Smirnov test yields a p-value greater than 0.05, the distribution is considered normal. Conversely, if p < 0.05, the distribution is deemed non-normal, and the skewness and kurtosis values will be examined. Variables with skewness and kurtosis values between -2 and +2 are considered to exhibit a normal distribution (George & Mallery, 2010).

The homogeneity of descriptive characteristics between groups will be tested using the chi-square test. For comparison of means between two independent groups, the independent samples t-test will be used if the data are normally distributed; otherwise, the Mann-Whitney U test will be applied. Changes within groups over repeated measurements will be analyzed using repeated measures ANOVA for normally distributed data, and the Friedman test for non-normally distributed data.

Ethical Considerations:

The study will commence following the receipt of ethical approval from the Koç University Ethics Committee and institutional permission from Koç University Hospital, where the research will be conducted. After obtaining the necessary permissions, informed consent will be secured from the patients using an "Informed Voluntary Consent Form," and subsequently, the survey forms will be distributed by the researcher. Written permission to use both scales in this study has been obtained via email from the respective authors.

References Abe, T., Matsuzaka, K., Nakayama, T., Otsuka, M., Sagara, A., Sato, F., Yumoto, T. (2021). Impact of air temperature and drug concentration on liquid emission from elastomeric pumps. Journal of Pharmaceutical Health Care and Sciences, 7(1), 1.

Arslan, M., Özdemir, L. (2015). Kemoterapiye bağlı gelişen bulantı-kusmanın yönetiminde kullanılan tamamlayıcı tedavi yöntemleri. Türk Onkoloji Dergisi, 30(2), 82-89.

Beck, A. T., Epstein, N., Brown, G., Steer, R. A. (1988). An inventory for measuring clinical anxiety: psychometric properties. Journal of Consulting and Clinical Psychology, 56(6), 893-897.

Burucu, R., Polat, H.T. (2024). Spiritual well-being levels and self-care agency of patients receiving chemotherapy with port catheter. Holistic Nursing Practice, 38(6), 331-340.

Can, A., Hintistan, S. (2021). Kemoterapi alan kanser hastalarının konfor düzeylerinin değerlendirilmesi. Bezmialem Science, 9(3), 310-316.

Chefchaouni, A.C., Ouedraogo, J-M., Bechar, H., Belahcen, M. J., Rahali, Y. (2023). Retrospective analysis of failures of ambulatory elastomeric pumps containing 5-FU in a hospital pharmacy unit. Journal of Oncology Pharmacy Practice, 29(1), 125-129.

Çıtlık, S.C., Çevik, S., Özden, G. (2018). Genel Konfor Ölçeği Kısa Formunun Türkçe geçerlik ve güvenirlik çalışması. Diyabet, Obezite ve Hipertansiyonda Hemşirelik Forumu, 10(2), 16-22.

Esfahani, H.M.D., Ghorbanpor, M.M.D., Tanasan, A.M.D. (2015), Implantable port devices, complications and outcome in pediatric cancer, a retrospective study. Iranian Journal of Pediatric Hematology and Oncology, 6(1), 1-8.

George, D., Mallery, M. (2010) SPSS for Windows Step by Step: A Simple Guide and Reference, 17.0 Update, 10th Edition, Pearson, Boston.

Gürlek, Ö., Yavuz, M. (2013). Cerrahi kliniklerde çalışan hemşirelerin ameliyat öncesi hasta eğitimi uygulama durumları. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 16(1), 8-15.

Hintistan, S., Pekmezci, H., Nural, N., Gülhan Güner, S. (2015). Kemoterapi Alan Hastalarda Psikolojik Semptomlar. Cumhuriyet Hemşirelik Dergisi, 4(1), 1-9.

Hou, Y. F., Zhao, A. P., Feng, Y. X., Cui, X. N., Wang, L. L., Wang, L. X. (2014). Nurses' knowledge and attitudes on comfort nursing care for hospitalized patients. International Journal of Nursing Practice, 20(6), 573-578.

International Agency for Research on Cancer (April 4, 2024). New report on global cancer burden in 2022 by world region and human development level. https://www.iarc.who.int/news-events/new-report-on-global-cancer-burden-in-2022-by-world-region-and-human-development-level/ Erişim Tarihi: 08.12.2024.

Kaykunoğlu, M., Tambağ, H. (2022). Ayaktan Kemoterapi Alan Hastaların Sosyal Destek ve Anksiyete Düzeylerinin Belirlenmesi. Celal Bayar Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi, 9(3), 429-435.

Kesici, S., Tuna, V., Özkan, S., Cengiz, E., Türkmen, A. (2017). Venöz port kateter implantasyonu uygulanan hastaların retrospektif analizi. Cukurova Medical Journal, 42, 604-605.

Kia, A., Waterson, J., Bargary, N., Rolt, S., Burke, K., Robertson, J., Garcia, S., Benavoli, A., Bergström, D. (2023). Determinants of intravenous infusion longevity and infusion failure via a nonlinear model analysis of smart pump event logs: Retrospective study. JMIR AI, 2, e48628.

Kim, K.S., Kwon, S.H. (2007). Comfort and quality of life of cancer patients. Asian Nursing Research, 1(2), 125-135.

Kolcaba, K., Schirm, V., Steiner, R. (2006). Effects of hand massage on comfort of nursing home residents. Geriatr Nurs. 27(2), 85-91.

Kutlu, R. (2015). Geçici/Kalıcı venöz kateterler ve port yerleştirme. Türk Radyoloji Derneği Semineri. İstanbul, Türkiye.

McCarthy, M., Glick, R., Green, J., Plummer, K., Peters, K., Johnsey, L., DeLuca, C. (2013). Comfort First: an evaluation of a procedural pain management programme for children with cancer. Psycho-Oncology, 22(4), 775-782.

Odabas, H., Ozdemir, N. Y., Ziraman, I., Aksoy, S., Abali, H., Oksuzoglu, B., Isik, M., Civelek, B., Dede, D., Zengin, N. (2014). Effect of port-care frequency on venous port catheter-related complications in cancer patients. International journal of clinical oncology, 19(4), 761-766.

Oran, N.T. (2009). Port kateter: Venöz yolu nasıl sürdürebiliriz? Maltepe Üniversitesi Hemşirelik Bilim ve Sanatı Dergisi. 2(3), 136-142.

Önder, H., Tekbaş, G., Turmak, M., İnal, A., Ekici, F., Gümüş, H, Önder, A. (2014). Image-guided subcutaneous port implantation in patients with malignant diseases. European Journal of General Medicine, 1, 1-6.

Özden, D., Çalıskan, N. (2012). Turkish nurses' level of knowledge regarding implantable port catheter care. Japan J Nurs Sci, 9, 1-8.

Öztaş, M., Alkan, İ., Öztaş, B. (2022). Determination of nursing practices regarding port catheter care. J Med Palliat Care, 3(1), 33-38.

Paiva, B.S.R., de Carvalho, A.L., Kolcaba, K., Paiva, C.E. (2015). Validation of the Holistic Comfort Questionnaire-caregiver in Portuguese-Brazil in a cohort of informal caregivers of palliative care cancer patients. Supportive Care in Cancer, 23(2), 343-351.

Paleczny, J., Banyś-Jafernik, B., Gazurek, K., Kierpieć, K., Szczerba, H., & Zipser, P. (2013). Long-term totally implantable venous access port systems--one center experience. Anaesthesiology Intensive Therapy, 45(4), 215-222.

Pinelli, F., Cecero, E., Degl'Innocenti, D., Selmi, V., Giua, R., Villa, G., Chelazzi, C., Romagnoli, S., & Pittiruti, M. (2018). Infection of totally implantable venous access devices: A review of the literature. Journal of Vascular Access, 19(3), 230-242.

Pu, Y. L., Li, Z. S., Zhi, X. X., Shi, Y. A., Meng, A. F., Cheng, F., Ali, A., Li, C., Fang, H., Wang, C. (2020). Complications and Costs of Peripherally Inserted Central Venous Catheters Compared With Implantable Port Catheters for Cancer Patients: A Meta-analysis. Cancer Nursing, 43(6), 455-467.

Sayin, Y., Aksoy, G. (2012). The effect of analgesic education on pain in patients undergoing breast surgery: within 24 hours after the operation. Journal of Clinical Nursing, 21(9-10), 1244-1253.

Sılgan, M. (2024). Kemoterapi Sırasında Dinletilen Müziğin Depresyon, Anksiyete, Stres Düzeyleri ve Kemoterapi Semptomlarına Etkisi. Yüksek Lisans Tezi, Maltepe Üniversitesi Lisansüstü Eğitim Enstitüsü, İstanbul, 2024.

Stewart, T., Pavlakis, N., Ward, M. (2010). Cardiotoxicity with 5-fluorouracil and capecitabine: more than just vasospastic angina. Intern Med J, 40, 303-307.

Shoemaker, L.K., Arora, U., Lima, C.M. (2004). 5-Fluoracil induced coronary vasospasm. Cancer Control, 11, 1-7.

Temiz, G., Durna, Z. (2020). Evaluation of quality of life and health care needs in cancer patients receiving chemotherapy. Journal of Cancer Education, 35(4), 796-807.

Turan, D., Cantürk, F. (2013). Kateter Uygulamaları ve Bakım Rehberi 2013. İstanbul: Sağlık Bakanlığı Tepecik Eğitim ve Araştırma Hastanesi Yayınları 2013.

Ulusoy, M., Şahin, N., Erkmen, H. (1998). Turkish version of The Beck Anxiety Inventory: Psychometric properties. Journal of Cognitive Psychother, 12, 28-35.

Uslu, Y., Olgun, N., Karanlık, H., User, İ. (2019). Port kateter uygulamaları: kanserli hastaların deneyimlerine ilişkin niteliksel bir çalışma. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi, 10(3), 464-472.

Yeşilbalkan, Ö.U. (2005). Onkoloji hastalarında sık kullanılan venöz giriş aracı impalante port kateter. C.Ü. Hemşirelik Yüksek Okulu Dergisi, 9(2), 49-54.

Yeşil, S., Tanyıldız, H.G., Ardıçlı, B., Tekgündüz, S.A., Çandır, M.O., Toprak, Ş., Bozkurt, C., Şahin, G. (2014). Santral venöz kateter komplikasyonları. Gazi Medical Journal, 25(4), 135-137.

Yilmaz, S.G., Arslan, S (2015). Effects of progressive relaxation exercises on anxiety and comfort of Turkish breast cancer patients receiving chemotherapy. Asian Pacific Journal of Cancer Prevention, 16(1), 217.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer,
* Able to understand Turkish and literate,
* Medically fit to participate in the study,
* Willing to participate in the study,
* Aged 18 years or older.

Exclusion Criteria:

* Diagnosed with a psychiatric disorder,
* Unable to communicate effectively,
* Refusing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 1 month
  The primary outcome measure of this study is the change in anxiety levels, as assessed by the Beck Anxiety Inventory (BAI), from baseline to one month post-intervention. This measure evaluates the effectiveness of the elastomeric pump education on reducing patient anxiety during chemotherapy treatment with 5-FU.

SECONDARY OUTCOMES:
Change in comfort levels from baseline to one month post-intervention, measured by the General Comfort Questionnaire-Short Form (GCQ-SF). | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Biruni University, Istanbul, Zeytinburnu
  - Biruni Üniversity, Istanbul

IPD SHARING:
Plan to Share IPD: No
Data will only be shared upon reasonable request and subject to approval by the ethics committee.